CLINICAL TRIAL: NCT05232019
Title: Association Between Embryo Implantation Rate and Maternal Age in Different Embryo Transplantation Cycles: a Retrospective Cohort Study
Brief Title: Association Between Embryo Implantation Rate and Maternal Age
Status: Completed | Type: Observational
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Principal Investigator of Reproductive Medicine Center of The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing University
Other Study IDs: SZ-2021-RIF
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile females: No less than 20 years old who were attending our clinical center for the first time were enlisted

SUMMARY:
To explore the relationship between maternal age and embryo implantation rate in patients undergoing assisted reproductive technology.

DETAILED DESCRIPTION:
The investigators designed a retrospective clinical trial conducted from January 2015 to December 2020 at the Reproductive Medicine Center of the Affiliated Drum Tower Hospital of Nanjing University Medical School. Infertility was defined as the failure of a clinical pregnancy after 12 months or more of regular unprotected intercourse with the same marriage partner. Patients experiencing infertility no younger than the age of 20 who attended the Reproductive Medicine Center of the Affiliated Drum Tower Hospital of Nanjing University Medical School for the first time and had experienced no less than one embryo transplantation between January 2015 and December 2019 were recruited. Patients who had experienced or canceled embryo transplantation cycles for any reason were excluded from this study. The gap year from December 2019 to December 2020 allowed researchers to follow up on the outcomes of pregnancies before 2020. Frozen cycles were performed when high-quality embryos existed to avoid unnecessary ovarian stimulation and oocyte retrieval processes. Investigators were blinded to the outcome of embryo transplantation, and information on pregnancy was gathered through telephone follow-up one year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. infertile patients
2. attended the Reproductive Medicine Center of the Affiliated Drum Tower Hospital of Nanjing University Medical School for the first time
3. had experienced no less than one embryo transplantation between January 2015 and December 2019

Exclusion Criteria:

canceled embryo transplantation cycles for any reason

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile females no less than 20 years old who were attending our clinical center for the first time were enlisted. In total, 17394 patients suffering from primary or secondary infertility were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 17394 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
embryo implantation rate | 60 days after embryo transplantation
  Fetal heartbeat can be visualized via ultrasound in order to definitely confirm the implantation of the embryo

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, PhD, Study Director — The affiliated Drum Towel Hospital of Nanjing University Medical School
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China